CLINICAL TRIAL: NCT07349030
Title: Data-driven Intervention to Reduce Pre-discharge Fall Risk After Stroke
Brief Title: Fall Risk Intervention for Stroke
Acronym: FRISKI
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: MGH Institute of Health Professions (Other)
Responsible Party: Principal Investigator, Prudence Plummer, Professor, MGH Institute of Health Professions
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 26AIREA1576341
Record Dates: First submitted 2025-12-29; First posted 2026-01-16 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Stroke
Keywords: falls; mobility; rehabilitation; physical therapy; physiotherapy; occupational therapy; speech language therapy
MeSH Terms: conditions — Stroke; Communication Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fall Prevention Rehabilitation (Experimental): In addition to usual care, participants randomized to the experimental intervention will receive 30-minute sessions of rehabilitation 6 times a week during the first week and 3 times a week thereafter until discharge. The intervention will target fall risk factors that are specific to the individual's fall risk profile at hospital admission. Patient and family education on fall prevention is also included.
  Interventions: Behavioral: Fall Prevention Intervention
- Dose-controlled Active Control (Active Comparator): In addition to usual care, participants randomized to the control intervention will receive 30-minute sessions of active control rehabilitation 6 times a week during the first week and 3 times a week thereafter until discharge. The intervention will be skilled rehabilitation that does not target known fall risk factors. Education on stroke recovery and stroke prevention will be provided as part of the control intervention.
  Interventions: Behavioral: Active Control

INTERVENTIONS:
Behavioral: Fall Prevention Intervention — The fall prevention rehabilitation program will be provided by a licensed physical therapist and will target modifiable fall risk factors known to be associated with future fall risk after inpatient rehabilitation for stroke. The intervention will be personalized to the individual's fall risk profile at admission. Participants will be educated about physical, cognitive/attentional, and environmental factors associated with falls.
  Arms: Fall Prevention Rehabilitation
Behavioral: Active Control — The control intervention will not include any of the key ingredients in the experimental intervention. The activities will not target known modifiable factors for fall risk, but the treatment will be a skilled therapy by a licensed provider, matching the dose of the experimental intervention. Participants in the control group will receive education about stroke, stroke recovery, stroke prevention, wellness, and community support groups.
  Arms: Dose-controlled Active Control

SUMMARY:
After stroke, falling is a common problem. Falls can lead to injury, as well as fear of future falls. It is important to try to prevent falls from happening after stroke. To goal of this study is to test a new treatment to try to prevent falls after stroke. The people in the study will be patients who are in the hospital receiving care after a stroke. While they are in the hospital, we will provide extra treatment that focuses on helping them not to fall. We will also teach the patients to understand risks for falls and how to avoid them. When they leave the hospital, we will send them a text message every day to ask if they have had any falls. Our goal is to see if patients who received the extra therapy have fewer falls than patients who did not receive the therapy and education to help avoid falls. If the extra treatment in the hospital can help stop people from falling after they leave the hospital, this will have a positive impact on their lives. By not falling, they will avoid the risk of injury and having to go back to the hospital. This project will help us know how we can help people with stroke live longer, healthier lives.

DETAILED DESCRIPTION:
Falls are one of the most significant problems for stroke survivors, often resulting in injury, fracture, rehospitalization, recurrent falls, fear of falling, avoidance of physical activity, and subsequent restricted social participation. The rate of falls among stroke survivors is exceptionally high, especially in the first 1-3 months after discharge home from the hospital. The high rate of early post-stroke falls occurs despite intensive inpatient rehabilitation and ongoing rehabilitation after hospital discharge. The central hypothesis to be tested in this study is that a personalized fall prevention intervention provided during inpatient rehabilitation will reduce fall risk before discharge compared to the control intervention (usual care plus dose-matched placebo activity) and reduce the 30-day and 90-day post-discharge fall rates. We will examine whether a targeted fall prevention intervention delivered during inpatient rehabilitation, in addition to usual care, can reduce fall risk classified by the clinical standard, Berg Balance Scale, at the time of discharge, more than usual care with dose-matched placebo activity (Aim 1). Upon admission to inpatient rehabilitation for stroke, patients without a prior history of falls who test positive for high fall risk using a validated, concise, bedside fall-risk assessment will be randomized 1:1 to experimental and control groups. We will compare differences between groups in the proportion that test positive for fall risk at discharge and the proportion who are discharged to a skilled nursing facility instead of home. Following hospital discharge, falls will be tracked via a daily text message survey for 90 days. We will compare the 30-day and 90-day fall rates between the experimental and control groups (Aim 2). There is a critical need to improve our rehabilitation practices for fall prevention early after stroke within current length-of-stay constraints. This study will determine whether an intensive, data-driven fall prevention intervention during inpatient rehabilitation can improve early post-stroke mobility and fall-related outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Inpatient rehabilitation admission for diagnosis of stroke
* Test positive for fall risk at admission (step-test and obstacle-test, "STOB", >/= 3 out of 8)
* No pre-stroke history of falls
* Community dwelling and independent in basic and instrumental activities of daily living prior to stroke
* Able to follow 1-step verbal command and demonstrate comprehension and decision-making capacity to consent to study participation
* Able to stand upright for 10 seconds with assistance of no more than one person

Exclusion Criteria:

* Brain hemorrhage due to trauma
* Prior stroke with residual physical or cognitive impairment
* Use of assistive device for ambulation prior to stroke
* Diagnosed with dementia
* Receptive or global aphasia
* Receiving chemotherapy in last 6 months or any cancer diagnosis with brain metastases

Ages: 45 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Estimated)
Dates: Start 2026-04-01 (Estimated); Primary Completion 2027-10-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Berg Balance Scale | Immediately post intervention
  Proportion of participants in each group who are at fall risk at hospital discharge, determined by the Berg Balance Scale (where fall risk is indicated by a score </= 43 out of 56).
Fall Rate | 30-days post intervention
  Prevalence of fallers (one or more falls) in each group 30 days after discharge
Fall Rate | 90 days post intervention
  Prevalence of fallers (one or more falls) in each group 90 days after discharge

SECONDARY OUTCOMES:
Functional Gait Assessment | Immediately post intervention
  Proportion of participants in each group who are at fall risk at discharge, determined by the Functional Gait Assessment (where fall risk is indicated by a score </= 13 out of 30).
Step-Obstacle Test | Immediately post intervention
  Proportion of participants in each group who are at fall risk at discharge, determined by the Step-Obstacle test combination (where fall risk is indicated by a score >/= 3 out of 8).
Discharge Disposition | Immediately post intervention
  Location discharged to from rehabilitation hospital

CONTACTS AND LOCATIONS:
Overall Officials: Prudence Plummer, PhD, Principal Investigator — MGH Institute of Health Professions
Locations (1):
- Spaulding Rehabilitation Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No